CLINICAL TRIAL: NCT02048059
Title: A Phase II, Open-Label, Multi-Center Study of ANG1005 in Breast Cancer Patients With Recurrent Brain Metastases
Brief Title: ANG1005 in Breast Cancer Patients With Recurrent Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Angiochem Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANG1005-CLN-04
Record Dates: First submitted 2014-01-21; First posted 2014-01-29 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer; Brain Metastases
Keywords: ANG1005; GRN1005; Low-density lipoprotein receptor-related protein (LRP-1); Targeted therapy; Breast cancer; Brain metastases; Brain tumor; Blood-brain barrier; Trastuzumab; Herceptin; Paclitaxel; Taxol; Breast cancer with brain metastases; Triple Negative; Triple negative breast cancer (TNBC); Herceptin 2 (HER2)-positive; HER2-negative; Metastatic brain tumors
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms; Triple Negative Breast Neoplasms | interventions — paclitaxel-Angiopep-2 conjugate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ANG1005 (Experimental): Participants received ANG1005 intravenously (IV) at a dose of 600 mg/m^2 on Day 1 of each 21-day cycle. ANG1005 will be administered for up to a maximum of one year, or until disease progression or adverse events (AE) that are not tolerated.
  Interventions: Drug: ANG1005

INTERVENTIONS:
Drug: ANG1005

SUMMARY:
This is a Phase 2 study to see if an investigational drug, ANG1005, can shrink tumor cells in breast cancer patients with recurrent brain metastases.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old
2. Breast cancer
3. Recurrent brain metastases from breast cancer
4. At least one radiologically-confirmed and measurable metastatic brain lesion ( ≥ 0.5 cm)
5. Neurologically stable
6. Karnofsky Performance Status (KPS) score ≥ 70
7. Adequate hematology and serum chemistry laboratory test results
8. Expected survival of ≥ 3 months

Exclusion Criteria:

1. Prior treatment with ANG1005/GRN1005
2. Evidence of symptomatic intracranial hemorrhage
3. Pregnancy or lactation
4. Inadequate bone marrow reserve
5. Any evidence of severe or uncontrolled diseases
6. Patients with the presence of an infection including abscess or fistulae, or known infection with hepatitis B or C or HIV
7. History of interstitial lung disease or evidence of clinically significant interstitial lung disease
8. Severe cardiac conduction disturbance
9. Central nervous system (CNS) disease requiring immediate neurosurgery intervention
10. Known severe hypersensitivity or allergy to paclitaxel or any of its components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Intracranial objective response rate (iORR) | Upon enrollment through end of study period (1 year after last patient is enrolled)

SECONDARY OUTCOMES:
Duration of intracranial objective response | Upon enrollment through end of study period (1 year after last patient is enrolled)
Median intracranial progression-free survival (PFS) | Upon enrollment through end of study period (1 year after last patient is enrolled)
Intracranial PFS rates at 3, 6 and 12 months | Upon enrollment through end of study period (1 year after last patient is enrolled)
6-month overall survival (OS) rate | Upon enrollment through end of study period (1 year after last patient is enrolled
Extracranial objective response rate (eORR) and duration of response | Upon enrollment through end of study period (1 year after last patient is enrolled
Number of Patients with adverse events | Upon enrollment through end of study period (1 year after last patient is enrolled
Plasma pharmacokinetics of ANG1005 | On Day 1 of Cycles 1 and 3
  To determine the drug concentration and distribution in the plasma. (AUC, Cmax, T1/2)
Intracranial ORR by modified Response Assessment in Neuro-Oncology (RANO) criteria | Upon enrollment through end of study period (1 year after last patient is enrolled)
Intracranial clinical benefit rate (iCBR) at 3 and 6 months | Upon enrollment through end of study period (1 year after last patient is enrolled)
Potential immunogenicity of ANG1005 | Upon enrollment through end of study period (1 year after last patient is enrolled)

CONTACTS AND LOCATIONS:
Overall Officials: Betty Lawrence, Study Director — Angiochem Inc
Locations (19):
- United States (19):
  - University of Arizona Cancer Center, Tucson, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California - LAC Medical Center, Los Angeles, California
  - University of Southern California - Norris Comprehensive Cancer Center, Los Angeles, California
  - UC - Irvine Chao Family Comprehensive Cancer Center, Orange, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - GRU Cancer Center - Georgia Regents University, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Maryland - Greenebaum Cancer Center, Baltimore, Maryland
  - National Cancer Institute, Bethesda, Maryland
  - Cancer & Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - The Long Islan Brain Tumor Center at Neurological Surgery P.C., Commack, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Univeristy of Texas Health Science Center in San Antonio, San Antonio, Texas

REFERENCES:
- See also: Safety, pharmacokinetics, and activity of GRN1005, a novel conjugate of angiopep-2, a peptide facilitating brain penetration, and paclitaxel, in patients with advanced solid tumors — http://www.ncbi.nlm.nih.gov/pubmed/22203732